CLINICAL TRIAL: NCT00193518
Title: A Phase II Trial Of Arsenic Trioxide (TRISENOX) In Patients With Relapsed Or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: Arsenic Trioxide in Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: CTI BioPharma (Industry)
Responsible Party: SCRI Oncology Research Consortium, SCRI
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LYM 33
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: Arsenic Trioxide

SUMMARY:
Additional active agents are needed to further improve the treatment of patients with CLL/SLL. Increasing information exists regarding the activity of arsenic trioxide in other hematologic malignancies. Since arsenic trioxide produces mild to moderate myelosuppression and is not as immunosuppressive as other available agents, it may be an additional treatment option for CLL/SLL. This study will evaluate the feasibility and toxicity of arsenic trioxide in patients with relapsed or refractory CLL/SLL

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will receive:

* Arsenic Trioxide

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Histologically proven B-cell CLL/SLL.
* Must have had a minimum of 1 and a maximum of 3 previous systemic regimens
* Must have progressive CLL/SLL
* Measurable or evaluable disease
* ECOG performance status 0, 1, or 2
* Age > 18 years.
* Patients with cytopenias caused by bone marrow involvement are eligible
* All patients must give written informed consent prior to entering this study.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Unstable active infection on the basis of neutropenia
* Previous severe opportunistic infections
* Severe immune mediated anemia or thrombocytopenia
* Serious underlying medical conditions
* Brain metastases or meningeal involvement
* History of other neoplasms
* Significant underlying heart dysfunction
* Women who are pregnant or

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41
Dates: Start 2004-04; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Progression-free survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States